CLINICAL TRIAL: NCT00811096
Title: Pilot Human Study of Tinidazole Efficacy For Radical Cure Of Plasmodium Vivax
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1477; HRPO Log#(A-15176);; Mahidol (TMEC 08-042)
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Malaria, Vivax
Keywords: Malaria, Vivax/*drug therapy; Tinidazole/pharmacology/*therapeutic use; Recurrence; Plasmodium vivax/*drug effects
MeSH Terms: conditions — Malaria, Vivax; Malaria; Recurrence | interventions — Tinidazole; Chloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Arm (Experimental)
  Interventions: Drug: Tinidazole
- Comparator Arm (Active Comparator): Comparator Arm
  Interventions: Drug: chloroquine

INTERVENTIONS:
Drug: Tinidazole — 2gms, p.o. q.d. for 5 days
  Arms: Treatment Arm
Drug: chloroquine
  Arms: Comparator Arm

SUMMARY:
Assess the efficacy of 2 grams of tinidazole given for 5 days with standard dose chloroquine to achieve radical cure of Plasmodium vivax within a 90 day follow-up period sufficient to justify an IND and formal phase II evaluation.

DETAILED DESCRIPTION:
This is a randomized, open-label study that will treat adult subjects with Plasmodium vivax infection with chloroquine for 3 days and tinidazole for 5 days concomitantly to assess efficacy for radical cure (clearance of blood and liver stages of infection). There will be randomization to a positive comparator arm treated with chloroquine and primaquine (definitive radical cure) in order to obtain an estimate of the rate of re-infection during the monitoring period in the study population.

A simple randomization procedure will assign subjects to one of the two arms (treatment arm or comparator arm). The ratio of assignment will be 2:1, treatment arm to the comparator arm. The exact number assigned to the treatment arm will vary depending on the initial outcome of early enrollees per the sequential analysis design of the trial. In the worse case scenario of no clear trend developing early, no more than 50 subjects will be required to complete the trial in the study drug arm in order to arrive at a conclusion regarding the study drug.

Follow-up period will be for 90 days. This will allow us to capture essentially all early relapses that would occur under normal circumstances, as well as assess if tinidazole may delay but not fully eliminate recurrence. Subjects without a recurrence at 90 days will be considered to have achieved radical cure.

This study will use a modified triangular test, a form of sequential analysis designed to enable repeated statistical analyses throughout the study recruitment period, while maintaining a pre-specified power and type I error. The trial can be stopped as soon as the information accumulated is considered sufficient to reach a conclusion and it will limit enrollment and exposure to a failing treatment regimen.

Results of this study will be sufficient to determine whether tinidazole should be designated as an "early kill" (an ineffective drug for vivax malaria radical cure with no future evaluation) or whether it is sufficiently efficacious to warrant further investment with an IND and formal phase II study to seek an SNDA.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and non-pregnant female volunteers that can communicate in the Burmese or Karen language.
* Age: Between 18 and 65 years (inclusive).
* Acute, symptomatic, blood smear positive diagnosis of Plasmodium vivax mono-infection.
* Ability to comprehend and comply with the requirements of the protocol.
* Willing to provide written informed consent.
* Willing to abstain from alcohol (EtOH) use during initial treatment and for 72 hours thereafter.
* Sexually active females must test negative on urine pregnancy test and must be counseled on an effective method of avoiding pregnancy (e.g., intrauterine contraceptive device; oral contraceptives; diaphragm or condom in combination with contraceptive jelly, cream or foam; Norplant® or Depo-Provera®), be surgically sterile, be post-menopause for at least one year, or be monogamous with a sterile sexual partner for at least 15 days prior to dosing with study product and at least 72 hours after their last dose of test drug.

Exclusion Criteria:

* Subjects positive for G6PD deficiency.
* Pregnant women (clinically or by positive urine β-HCG) and nursing mothers.
* Concomitant use of metronidazole, albendazole or mebendazole.
* Any malaria treatment or use of azithromycin or other macrolides, tetracyclines, sulfonamides, doxycycline, tetracycline or other sulfa based or other drug with antimalarial activity for the previous 4 weeks prior to screening. Additionally, concomitant use of phenobarbitol, rifampin, phenytoin, fosphenytoin, cimetidine, ketoconazole, cholestryramine constitute exclusion criteria.
* Significant health problems, including, but not limited to significant, cardiac, renal or liver disease or lab abnormalities and those subjects in whom it is suspected that they will not abstain from alcohol use during treatment and for the subsequent 3 days.
* Mixed malaria infection on admission determined by malaria smear and/or any positive HRP2 antigen testing.
* A previous history of significant intolerance or hypersensitivity to the study drug tinidazole or to chloroquine or primaquine. (nausea alone from previous primaquine use will not be an excluding factor unless subject was unable to complete a primaquine course due to this discomfort.)
* Subjects that have received transfusions within the previous 30 days.
* Presenting hematocrit <25%.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-11; Primary Completion 2009-01 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Cure is defined as absence of malaria infection on thick/thin malaria smears up to and on day 63 after initial clearance of parasitemia. Subjects will be followed to day 90 to rule out delayed presentation of malaria (as opposed to cure). | 63 days

SECONDARY OUTCOMES:
Recurrence (relapse, recrudescence or re-infection) of Plasmodium vivax between blood stage clearance and 90 days. | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Francois Nosten, MD, Principal Investigator — Malaria Research Unit, Thailand
Locations (1):
- Malaria Research Unit, 68/30 Ban Toong Road, P.O. Box 46, Mae Sot, Changwat Tak, Thailand

REFERENCES:
- [Derived] Macareo L, Lwin KM, Cheah PY, Yuentrakul P, Miller RS, Nosten F. Triangular test design to evaluate tinidazole in the prevention of Plasmodium vivax relapse. Malar J. 2013 May 29;12:173. doi: 10.1186/1475-2875-12-173. PMID 23718705